CLINICAL TRIAL: NCT01070251
Title: Effects of a Multimodal Preference-based Parental Intervention on Preschoolers' Physical Activity Behaviour - a Cluster-randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Joachim E. Fischer, Professor >Dr. med. MSc, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CRTLasti_PA_kiga
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Existing state-sponsored PA program (Active Comparator): standard children-focused gym lessons approach
  Interventions: Behavioral: State-sponsored PA program
- Participatory intervention plus state-sponsored PA program (Active Comparator): Participatory parent-focused intervention over nine months in addition to state-sponsored PA program
  Interventions: Behavioral: Participatory parent-focused intervention; Behavioral: State-sponsored PA program

INTERVENTIONS:
Behavioral: Participatory parent-focused intervention — Parent workshops and internet-based support to establish healthy physical activity routines, added to existing state-sponsored PA program
  Other Names: "Ene mene fit - Eltern machen mit!"
  Arms: Participatory intervention plus state-sponsored PA program
Behavioral: State-sponsored PA program — Preschool children receive twice a week 60 minutes of physical activity lessons over 6 months by an external gym trainer
  Other Names: Standard physical activity lessons

SUMMARY:
This study investigates whether a preschool-based physical activity intervention involving parents as active agents of behavioral change affects objectively measured physical activity in preschool children.

DETAILED DESCRIPTION:
In the last 25 years, obesity in children has increased dramatically in Germany (Lampert et al. 2007, Stolzenberg et al., 2007) and other western societies. Lack of physical activity (PA) is one important factor contributing to obesity development. However, healthy behaviors are established early in life (adiposity rebound: Reilly 2008), which underlines the importance of early interventions. Preschools therefore might be an ideal setting for interventions to promote physical activity. While previous preschool interventions were directly aimed at the children's physical activity behaviors (e.g. promoting activity by sports lessons), parents as influential caregivers were mainly involved in educational ways and by information (e.g. newsletters, physical activity homework).

The current intervention takes a participatory approach to involve parents as active agents of behavioral change. The study aim is to evaluate the effects of the participatory preference-based parental intervention on preschoolers' objectively measured physical activity behaviour and Body Mass Index (BMI). The intervention can easily be added as a parent module to existing children-focused physical activity programmes.

In several workshops, parents are presented a set of possible project ideas for improving everyday physical activity in the preschools. After forming teams, they either select project ideas from the preexisting menu or develop ideas de novo and then implement them into the local preschool environment.

The intervention is implemented in the frame of an existing state-sponsored physical activity (PA) program offering twice weekly sports lessons by external gym trainers to preschoolers over a period of 6 months. Preschools in the control arm get the state-sponsored PA program only. Preschools in the intervention arm get the participatory parent-focused PA intervention in addition to the existing state-sponsored PA program.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* Participation in the standard physical activity lesson twice weekly

Exclusion Criteria:

* Age under 3 years or above 6 years
* Serious atopic dermatitis
* Genetic conditions
* Metabolic diseases
* Acute infectious diseases

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 826 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change in physical activity as measured by accelerometry and heart rate | 0,6 and 12 months
  before intervention (0 months), 6 and 12 months later

SECONDARY OUTCOMES:
Change in Body Mass Index, percent fat mass (based on skin folds), waist-to-height ratio and waist circumference Change in blood pressure, sympathetic/parasympathetic tone. Sleep quantity by accelerometry. | 0, 6 and 12 months
  before intervention (0 months), 6 and 12 months later

OTHER OUTCOMES:
Change in quality of life and subjective wellbeing | 0, 6 and 12 months
  before intervention (0 months), 6 and 12 months later

CONTACTS AND LOCATIONS:
Overall Officials: Joachim E Fischer, Prof MD MSc, Study Director — Mannheim Insitute of Public Health, Mannheim Medical Faculty, Heidelberg University
Locations (2):
- Germany (2):
  - Mannheim Institute of Public Health, University of Heidelberg, Mannheim, Baden-Wurttemberg
  - Mannheim Institute of Public Health, Mannheim, Baden-Wurttemberg

REFERENCES:
- [Background] Reilly JJ, Kelly L, Montgomery C, Williamson A, Fisher A, McColl JH, Lo Conte R, Paton JY, Grant S. Physical activity to prevent obesity in young children: cluster randomised controlled trial. BMJ. 2006 Nov 18;333(7577):1041. doi: 10.1136/bmj.38979.623773.55. Epub 2006 Oct 6. PMID 17028105
- [Background] Taylor RW, Mcauley KA, Williams SM, Barbezat W, Nielsen G, Mann JI. Reducing weight gain in children through enhancing physical activity and nutrition: the APPLE project. Int J Pediatr Obes. 2006;1(3):146-52. doi: 10.1080/17477160600881247. PMID 17899632